CLINICAL TRIAL: NCT05238714
Title: An Open-label Study of Excretion Balance and Pharmacokinetics Following a Single Oral Dose of [14C]-Venglustat (2.67 MBq) in Healthy Male Subjects
Brief Title: Excretion Balance, Pharmacokinetics, and Metabolism Following of [14C]-Venglustat Administration in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BEX13673; 2019-001041-41 (EudraCT Number); U1111-1180-5557 (Registry Identifier: ICTRP)
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Disorders of Sphingolipid Metabolism; Healthy Volunteers
MeSH Terms: interventions — venglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [14C] venglustat (Experimental): Single dose of [14C] venglustat Oral Solution under fasting conditions
  Interventions: Drug: venglustat

INTERVENTIONS:
Drug: venglustat — Powder for Oral solution

SUMMARY:
Primary Objectives:

* To determine the excretion balance and systemic exposure of radioactivity after oral administration of [14C]-venglustat.
* To determine the pharmacokinetics (PK) of venglustat and its contribution to the overall exposure of radioactivity.
* To determine the metabolic pathways, metabolite profile, chemical structures and main excretion route of the main venglustat metabolites and the metabolite contribution to the overall exposure of radioactivity.

Secondary Objective:

To assess the clinical and biological tolerability of oral solution of venglustat

DETAILED DESCRIPTION:
43 days

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 50.0 and 100.0 kg, inclusive, body Mass Index 18 to 32 kg/m2, inclusive
* Certified as healthy by a comprehensive clinical assessment
* Normal vital signs after 10 minutes resting in supine position
* Standard 12-lead electrocardiogram (ECG) parameters after 10 minutes resting in supine position in the following ranges; 120 ms≤PR≤230 msec, QRS≤120 msec, QTc≤450 msec and normal ECG tracing unless the Investigator considers an ECG tracing abnormality to be not clinically relevant
* Laboratory parameters within the normal range
* Having given written informed consent prior to undertaking any study-related procedure
* Covered by a health insurance system where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research
* Not under any administrative or legal supervision
* Normal renal function as expressed by a creatinine clearance >80 mL/min as calculated by the Cockroft and Gault formula
* Male subjects who agree to use condoms, whose female partner(s) are of childbearing potential (including lactating women), must accept to use, during sexual intercourse, a double contraception method (unless they underwent surgical sterilization) until 90 days after the end of study

Exclusion Criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness
* Frequent headaches and/or migraine, recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* Blood donation, any volume, within 3 months before inclusion.
* Symptomatic postural hypotension, irrespective of the decrease in blood pressure.
* Presence or history of clinically significant drug hypersensitivity, or allergic disease diagnosed and treated by a physician that in the opinion of the Investigator would compromise subject safety.
* History or presence of drug or alcohol abuse (alcohol consumption more than 14 units per week on a regular basis) in the 5 years prior to screening.
* Smoking or using nicotine replacement products or e-cigarettes regularly more than 5 cigarettes or equivalent per week, unable to stop smoking during the study (occasional smoker can be enrolled).
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day)
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication; any vaccination or any medications known to be CYP3A4 inducers within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the Investigator at screening.
* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.
* Any subject enrolled in or having participated, in [this or] any other clinical study involving an investigational medicinal product (IMP) according to applicable regulations/guidelines in the 3 months prior to dosing of this study.
* Any subject who cannot be contacted in case of emergency.
* Any subject who is the Investigator or any sub investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
* Confirmed positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, tricyclic antidepressants, opiates including methadone).
* Positive alcohol breath test
* Any subject with specific dietary habits, such as vegan.
* Any subject with irregular bowel habits (more than 3 bowel movements/day or less than 1 every 2 days).
* Any subject undergoing dental care or presenting with dental caries.
* Any subject who is occupationally exposed to radiation as defined in the Ionizing Radiations Regulations 2017
* Participation in a trial with 14C-radiolabelled medication in the 12 months preceding the study.
* Radiation exposure, including that from the present study and radiopharmaceuticals or radionuclides in therapeutic or diagnostic procedures, but excluding background radiation, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years.
* Any consumption of citrus (grapefruit, orange, etc) or their juices within 5 days before inclusion

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Percentage of radioactive dose excreted in urine and faeces | Day -1 up to max Day 43
  Percentage of radioactive dose excreted in urine and faeces
Cmax of plasma and blood radioactivity | Day 1 up to max Day 43
  Maximum plasma or blood concentration observed
AUC Last of plasma and blood radioactivity | Day 1 up to max Day 43
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time, tlast (time corresponding to the last concentration above the limit of quantification, Clast)
AUC Last of plasma venglustat | Day 1 up to max Day 43
tmax of plasma and blood radioactivity | Day 1 up to max Day 43
  Time to Cmax
tmax of plasma venglustat | Day 1 up to max Day 43
  Time to reach Cmax

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Day 1 up to max Day 43
  Number of participants with AEs
Percentage of venglustat metabolites in plasma | Day 1 up to max Day 43
  Percentage of venglustat metabolites in plasma
Percentage of venglustat metabolites in urine | Day 1 up to max Day 43
  Percentage of venglustat metabolites in urine
Percentage of venglustat metabolites in faeces | Day 1 up to max Day 43
  Percentage of venglustat metabolites in faeces

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number :8260001, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: BEX13673 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25220&tenant=MT_SNY_9011